CLINICAL TRIAL: NCT06957678
Title: Artificial Intelligence-Based Prediction of Lymph Node Metastasis and Nodal Station Involvement in Gastric Cancer Using Preoperative Multimodal Imaging and Pathology Data
Brief Title: AI-Based Prediction of Lymph Node Metastasis in Gastric Cancer Using Preoperative Multimodal Data
Status: Enrolling by invitation | Type: Observational
Sponsor: Qun Zhao (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Nanjing University School of Medicine (Other); Baoding First Central Hospital (Other); Hengshui People's Hospital (Other); No.1 Hospital of Shijiazhuang City (Unknown); The Second Affiliated Hospital of Xingtai Medical College (Unknown)
Responsible Party: Sponsor-Investigator, Qun Zhao, Professor, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: GC-RAD-AI-2025-02
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer Adenocarcinoma Metastatic; Lymph Node Metastasis; Artificial Intelligence (AI) in Diagnosis
MeSH Terms: conditions — Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence-Based Predictive Model for Lymph Node Metastasis — The intervention is an artificial intelligence-based predictive model developed using preoperative multimodal data, including contrast-enhanced CT images, preoperative histopathological findings, and clinical features. The model is designed to predict (1) the presence or absence of lymph node metastasis, (2) the specific lymph node stations involved, and (3) the individual lymph nodes involved. Each lymph node's metastatic status is confirmed by serial pathological sectioning of surgically retrieved nodes, ensuring a highly accurate reference standard for model training and validation. This distinguishes the intervention from traditional imaging-based assessments and from other AI models that do not use individually validated lymph node pathology.

SUMMARY:
This study aims to develop and validate an artificial intelligence (AI) system that can predict whether lymph node metastasis has occurred in patients with gastric cancer before surgery. Using preoperative imaging and pathology data, the AI models will not only predict if metastasis is present but also identify which specific lymph node stations or individual lymph nodes are involved. All lymph nodes will be carefully removed during surgery and examined one by one with detailed pathological methods to ensure accurate diagnosis. The goal is to improve the accuracy of lymph node assessment and assist doctors in making better treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older

Histologically confirmed gastric adenocarcinoma

Scheduled for curative-intent gastrectomy with lymphadenectomy

Completed preoperative imaging with contrast-enhanced CT or MRI

Available preoperative biopsy pathology report

Able and willing to provide written informed consent

Exclusion Criteria:

* Evidence of distant metastasis on preoperative imaging

Prior chemotherapy, radiotherapy, or major abdominal surgery

Severe comorbidities contraindicating surgery

Incomplete or poor-quality preoperative imaging or pathology data

Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult patients diagnosed with gastric adenocarcinoma who are scheduled to undergo curative-intent gastrectomy with lymphadenectomy. Participants must have completed preoperative imaging studies and histopathological evaluation. All enrolled patients will have individually retrieved lymph nodes evaluated by detailed pathological examination to provide a definitive reference for lymph node metastasis status.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the AI Model in Predicting Presence of Lymph Node Metastasis in Gastric Cancer | From Preoperative Evaluation to Completion of Postoperative Pathological Analysis (Approximately 4-6 Weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Hospital of Hebei Medical University, Shijiazhuang, None Selected, China